CLINICAL TRIAL: NCT01951040
Title: Effect of Oxytocin Administered During Labor on the Onset and Duration of Breastfeeding: A Retrospective Cohort Study.
Brief Title: Effect of Synthetic Oxytocin Administered During Labor on Breastfeedings
Status: Completed | Type: Observational
Sponsor: Hospital Materno-Infantil de Málaga (Other)
Responsible Party: Principal Investigator, Ernesto González Mesa, PHD Obstetrics and Gynecology, Hospital Materno-Infantil de Málaga
Other Study IDs: OXYTO-2011-BRSTF
Record Dates: First submitted 2013-09-19; First posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Breastfeeding
Keywords: Oxytocin, breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Oxytocin: Oxytocin was administered during labor
- No Oxytocin: Oxytocine was not administered during labor

SUMMARY:
This study was designed as a retrospective cohort study where patients given synthetic oxytocin during labor induction were considered as the exposed cohort, and patients not given oxytocin formed the non-exposed cohort. Four hundred of the 7465 children born at our maternity during 2006 were randomly selected. Information about breast-feeding was available for 316 of these children. Eventual confounding or adjustment factors were analyzed using stratified and multivariate analysis (logistic regression

DETAILED DESCRIPTION:
Study population consisted of children born in our center (Hospital Materno-Infantil in Malaga) during 2006. Our hospital is a tertiary center of the Spanish national health system where were born 7465 children, representing 41.2% of all babies born in our province, from 7246 deliveries during that year 21. Random sample size was estimated at 400, with a 95% confidence levels and a 20% power, considering an expected RR of 0.82 22, a ratio between exposed and unexposed groups of 1.5, and a 20% loss. The sample selection was done by random sampling with the SPSS random number generator.

Once approval was obtained from the ethics and research committee of the hospital, recruitment and monitoring of selected cases was started during 2011. Data were collected by review of clinical records and interviews with the mothers (particularly to record breast-feeding type and duration). Patients were referred to the hospital for a semi-structured interview in which data were collected for type and duration of feeding. Clinical records were used as information sources for obstetric variables. Both the interviews and the review of medical records were blinded and conducted by the study authors in different days

ELIGIBILITY:
Inclusion Criteria:

* children born in our center (Hospital Materno-Infantil in Malaga) during 2006

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population consisted of children born in our center (Hospital Materno-Infantil in Malaga) during 2006. Our hospital is a tertiary center of the Spanish national health system where were born 7465 children, representing 41.2% of all babies born in our province, from 7246 deliveries during that year
Sampling Method: Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2011-02; Primary Completion 2013-01 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
use of breast-feeding | 21 months. From March 2011 to december 2012
  both, alone and combined with bottle feeding

SECONDARY OUTCOMES:
duration of breastfeeding | 21 months. From March 2011 to december 2012
  Number of months

CONTACTS AND LOCATIONS:
Overall Officials: ERNESTO GONZÁLEZ-MESA, PHD, Principal Investigator — Hospital Materno-Infantil de Málaga

REFERENCES:
- [Derived] Garcia-Fortea P, Gonzalez-Mesa E, Blasco M, Cazorla O, Delgado-Rios M, Gonzalez-Valenzuela MJ. Oxytocin administered during labor and breast-feeding: a retrospective cohort study. J Matern Fetal Neonatal Med. 2014 Oct;27(15):1598-603. doi: 10.3109/14767058.2013.871255. Epub 2014 Jan 13. PMID 24289796